CLINICAL TRIAL: NCT01189071
Title: Preoperative Use of Darifenacin (Enablex) to Alleviate Postoperative Ureteral Stent Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Co-Investigator left institution. No data analysis occurred.
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB 1119697
Record Dates: First submitted 2010-08-19; First posted 2010-08-26 (Estimated); Results first posted 2016-11-21 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Overactive Bladder; Renal Colic; Pain, Postoperative
Keywords: Stents [E07.695.750]; Darifenacin (C101207); Kidney calculi
MeSH Terms: conditions — Urinary Bladder, Overactive; Renal Colic; Pain, Postoperative; Kidney Calculi | interventions — darifenacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Darifenacin (Active Comparator): 3 days of preoperative darifenacin anticholinergic medication
  Interventions: Drug: Darifenacin
- no pill (No Intervention): The control group will have the standard of care which is no preoperative anticholinegic medication.

INTERVENTIONS:
Drug: Darifenacin — an M3 selective anticholinergic medication. M3 muscarinic receptors are felt to be related to bladder and ureteral contractility. The ureteral and bladder spasms related to ureteral stents are felt to be due to inappropriate contractions. By using a selective M3 receptor, it is felt that there will be fewer side effects. Participants will be placed on the standard 15 mg oral daily dosage for 3 days prior to the stent being placed, day 3 being the am of the surgery.
  Other Names: Enablex
  Arms: Darifenacin

SUMMARY:
This will be a randomized two arm prospective study to evaluate postoperative ureteral stent pain. One arm will be given 3 days of preoperative darifenacin and the control group will have the standard of care which is no preoperative anticholinergic medication. The primary endpoints will be decreased pain scores and less ER visits and hospital admissions for stent difficulty. These will be assessed by a pain diary completed by the participant as well as a questionnaire when the participant returns to clinic for stent removal. Also included in evaluation of the primary end point will be patient phone calls, ER visits and admissions for stent difficulty. Secondary endpoints will be narcotic and postoperative anticholinergic use. This will also be assessed with the pain diary completed by the participant. Participants will be included in the study if they are undergoing a procedure that a stent will likely be required. This will include participants who will have ureteroscopy or extracorporeal shock wave lithotripsy and a stone 1 cm or larger. Also participants with stones smaller than 1 cm who due to anatomy of the ureter or kidney will likely need a stent on preoperative evaluation will also be included in the study. Included as well in the study are participants who will undergo renal or ureteral surgery that a ureteral stent will be utilized. Participants will be randomized after consent is obtained into two groups. One group will receive standard of care which is no preoperative anticholinergic medications. The second group will receive the three day treatment with darifenacin pre procedure. Participants in the second group will be instructed on side effects of darifenacin and given appropriate contact information prior to initiation of the medication. Both groups will be followed postoperatively with a pain diary. Postoperative follow up will continue until the stent is removed 1-2 weeks after the procedure. The exact time of stent removal will depend on the success and nature of the surgery and will be at the discretion of the surgeon. Participants will be able to voluntarily stop the medication for any reason as well as if they have serious side effects from the medication. Data to be collected from each group includes age, gender, race, prior ureteral stents, prior renal or ureteral surgery, past medical history, allergies, current medications and urinary complaints.

DETAILED DESCRIPTION:
The purpose of the study is to determine if preoperative dosing of darifenacin will assist in postoperative ureteral stent pain. This will be a randomized two arm prospective study to evaluate postoperative ureteral stent pain. One arm will be given 3 days of preoperative darifenacin and the control group will have the standard of care which is no preoperative anticholinergic medication. The primary endpoints will be decreased pain scores and less ER visits and hospital admissions for stent difficulty. These will be assessed by a pain diary completed by the participant as well as a questionnaire when the participant returns to clinic for stent removal. Also included in evaluation of the primary end point will be patient phone calls, ER visits and admissions for stent difficulty. Secondary endpoints will be narcotic and postoperative anticholinergic use. This will also be assessed with the pain diary completed by the participant. Participants will be included in the study if they are undergoing a procedure that a stent will likely be required. This will include participants who will have ureteroscopy or extracorporeal shock wave lithotripsy and a stone 1 cm or larger. Also participants with stones smaller than 1 cm who due to anatomy of the ureter or kidney will likely need a stent on preoperative evaluation will also be included in the study. Included as well in the study are participants who will undergo renal or ureteral surgery that a ureteral stent will be utilized. Participants will be randomized after consent is obtained into two groups. One group will receive standard of care which is no preoperative anticholinegic medications. The second group will receive the three day treatment with darifenacin pre procedure. Participants in the second group will be instructed on side effects of darifenacin and given appropriate contact information prior to initiation of the medication. Both groups will be followed postoperatively with a pain diary. Postoperative follow up will continue until the stent is removed 1-2 weeks after the procedure. The exact time of stent removal will depend on the success and nature of the surgery and will be at the discretion of the surgeon. Participants will be able to voluntarily stop the medication for any reason as well as if they have serious side effects from the medication. Data to be collected from each group includes age, gender, race, prior ureteral stents, prior renal or ureteral surgery, past medical history, allergies, current medications and urinary complaints.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be included in the study if they are undergoing a procedure that a stent will likely be required. This will include participants who will have ureteroscopy or extracorporeal shock wave lithotripsy and a stone 1 cm or larger.
* Also participants with stones smaller than 1 cm who due to anatomy of the ureter or kidney will likely need a stent on preoperative evaluation will also be included in the study.
* Included as well in the study are participants who will undergo renal or ureteral surgery that a ureteral stent will be utilized.

Exclusion Criteria:

* Those who do not meet inclusion criteria-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-08; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark R Wakefield, MD, Principal Investigator — University of Missouri Healthcare, USA
Locations (1):
- University of Missouri Healthcare, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three participants were recruited to the study, but no data were collected or analyzed as the author of the study left the institution and the study was terminated.
Period: Overall Study
Arm/Group | Darifenacin | no Pill
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Three participants were recruited to the study, but no data were collected or analyzed as the author of the study left the institution and the study was terminated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Darifenacin | no Pill | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
  <=18 years |  |  | 0
  Between 18 and 65 years |  |  | 0
  >=65 years |  |  | 0
Gender
  Female |  |  | 0
  Male |  |  | 0
Region of Enrollment
  United States |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Decreased Post Operative Ureteral Stent Pain, Evidenced by Decreased Pain Scores, Less ER Visits/Hospital Admits, or Patient Phone Calls for Stent Pain/Difficulty
Description: Decreased post operative ureteral stent pain, evidenced by decreased pain scores, less ER visits/hospital admits, or patient phone calls for stent pain/difficulty, as compared to the "standard of care" patient with no preop Darifenacin
Time Frame: 24 months
Population: as for baseline characteristics
Arm/Group | Darifenacin | no Pill
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Decreased Use of Narcotic and Anticholinergic Medication Use Postoperatively.
Description: Decreased use of narcotic and anticholinergic medication use postoperatively, compared to the "standard of care" patient
Time Frame: end of study with 30 patients recruited
Population: as for baseline characteristics
Arm/Group | Darifenacin | no Pill
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Darifenacin | no Pill
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Three participants were recruited to the study, but no data were collected or analyzed as the author of the study left the institution and the study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes